CLINICAL TRIAL: NCT00035932
Title: Phase III Open Label Atazanavir (BMS-232632) in Combination With Ritonavir or Saquinavir, and Lopinavir/Ritonavir, Each With Tenofovir and a Nucleoside in Subjects With HIV
Brief Title: Atazanavir (BMS-232632) in Combination With Ritonavir or Saquinavir, and Lopinavir/Ritonavir, Each With Tenofovir and a Nucleoside in Subjects With HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI424-045; NCT00028054 (obsolete NCT alias)
Expanded Access: Available
Record Dates: First submitted 2002-05-06; First posted 2002-05-08 (Estimated); Results first posted 2010-12-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; Tenofovir; Nucleosides; Saquinavir; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- I (Active Comparator): ATV 300 mg + RTV 100 mg + TDF 300 mg + nucleoside of choice
  ATV , RTV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
  Interventions: Drug: Atazanavir + ritonavir + tenofovir + nucleoside
- II (Active Comparator): ATV 400 mg + SQV 1200 mg + TDF 300 mg + nucleoside of choice
  ATV, SQV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
  Interventions: Drug: Atazanavir + saquinavir + tenofovir + nucleoside
- III (Active Comparator): LPV/RTV 400/100 mg + TDF 300 mg + nucleoside of choice
  LPV/RTV twice daily, TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
  Interventions: Drug: Lopinavir/ritonavir + tenofovir + nucleoside

INTERVENTIONS:
Drug: Atazanavir + ritonavir + tenofovir + nucleoside — Active Comparator, Capsules, tablets, Oral
  Other Names: BMS-232632; Reyataz
  Arms: I
Drug: Atazanavir + saquinavir + tenofovir + nucleoside — Active Comparator, Capsules, tablets, Oral
  Other Names: BMS-232632; Reyataz
  Arms: II
Drug: Lopinavir/ritonavir + tenofovir + nucleoside — Active Comparator, Capsules, tablets, Oral
  Arms: III

SUMMARY:
The purpose of this study is to learn how well atazanavir (ATV) works in combination with ritonavir (RTV) or saquinavir (SQV) with tenofovir (TDF) and a nucleoside to reduce the viral load of treatment experienced subjects with human immunodeficiency virus (HIV). There is a comparison arm with lopinavir (LPV)/RTV and TDF and a nucleoside.

ELIGIBILITY:
Inclusion Criteria:

* Virologic failure to 2 or more highly active antiretroviral therapy (HAART) regimens that, in total, have included at least one drug from all approved classes protease inhibitors, non-nucleoside reverse transcriptase inhibitors, nucleoside reverse transcriptase inhibitors (PI, NNRTI, NRTI):

  1. Currently on a failing HAART regimen with 2 qualifying plasma viral load measurements (hospital/clinic value within 4 weeks of screening with viral load equivalent to =>1,000 c/mL on the Roche Amplicor[TM] and central lab measurements of =>1,000 c/mL (Roche Amplicor[TM]) within 4 weeks of randomization
  2. Cluster of Differentiation 4 (CD4) cell count =>50 cells/mm3 obtained within 4 weeks prior to randomization
* =>16 years of age (or minimum age as determined by local regulations or as legal requirements dictate);
* History of prior virologic response to at least one HAART regimen, defined as a 1.0 log10 decline or a decline in viral load to <400 c/mL by Roche Amplicor or <500 c/mL by Chiron Quantiplex branched DNA (bDNA) assay
* Both females of child bearing potential and males must utilize effective barrier contraception to reduce transmission of sexually transmitted disease, including human immunodeficiency virus (HIV). Other contraception in addition to barrier methods is permitted; interaction between atazanavir and oral contraceptives has not been studied.
* Subjects must be able to provide written informed consent;
* Subjects should be available for follow-up for a period of at least 48 weeks
* Baseline laboratory values measured within 2 weeks prior to initiating study drugs as follows:

  1. serum creatine <1.5 times the upper limit of normal (ULN)
  2. total serum lipase <1.4 times the ULN
  3. liver enzymes alanine aminotransferase (AST), aspartate aminotransferase (ALT) <3 times the ULN
  4. total serum bilirubin <1.5 times the ULN

Exclusion Criteria:

* Prior use (=>3 days) of atazanavir, TVF or LPV/RTV; if history of SQV, then must be phenotypically sensitive
* the current failing antiretroviral regimen must have been administered for at least eight weeks at he initiation of screening and must not include both a PI and NNRTI
* Presence of a newly diagnosed HIV-related opportunistic infection or any medical requiring acute therapy at the time of enrollment
* Proven or suspected acute hepatitis in the 30 days prior to study entry. Subjects with chronic hepatitis are eligible provided that their liver function enzymes (ALT/AST) are <3 x ULN
* Previous therapy with agents with significant systemic myelosuppressive, neurotoxic, pancreatoxic, hepatoxic or cytotoxic potential within 3 months of study start or the expected need for such therapy at the time of enrollment of therapy with methadone or ribavirin/interferons or treatment with neurotoxic drugs or drugs that affect Cytochrome P450 3A4 (CYP3A4).
* Active alcohol or substance use sufficient, in the Investigator's opinion, to prevent adequate compliance with study therapy or to increase the risk of developing pancreatitis or chemical hepatitis
* Intractable diarrhea (=> 6 loose stools/day for at least 7 days consecutive days) within 30 days prior to study entry
* Pregnancy or breast-feeding
* History of hemophilia
* Presence of cardiomyopathy
* Any one of the following:

  1. Heart rate-corrected QT (QTc) interval >450 msec on the screening electrocardiogram (EKG)
  2. Heart rate <40 beats per minute (bpm)
  3. Pause length >3 seconds seen on EKG
  4. Clinical symptoms potentially related to heart block
  5. Third degree heart block
* History of acute or chronic pancreatitis
* If choosing 2'-3' dideoxyinosine (ddI) or 2',3'-didehydro-3'-deoxythymidine (d4T) as the NRTI: History or signs and symptoms of bilateral peripheral neuropathy => Grade 2 at the time of screening
* Inability to tolerate oral medications
* Any other clinical conditions or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for study or unable to comply with the dosing requirements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2001-11; Primary Completion 2003-07 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- United States (26):
  - San Francisco, California
  - Torrance, California
  - Boulder, Colorado
  - Altamonte Springs, Florida
  - Fort Lauderdale, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Decatur, Georgia
  - Honolulu, Hawaii
  - Boise, Indiana
  - Wichita, Kansas
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Brookline, Massachusetts
  - Fall River, Massachusetts
  - East Orange, New Jersey
  - Newark, New Jersey
  - Buffalo, New York
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Dallas, Texas
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 571 human immunodeficiency virus (HIV)-infected participants were enrolled; 358 (63%) were randomized to treatment. Of the 213 not randomized, 194 did not meet eligibility criteria; other reasons include duplicate enrollment (4), accrual closed (1), noncompliance (1), serious adverse event (2), patient request (11), missing information (4).
Groups:
- ATV 300 mg / RTV: atazanavir (ATV) 300 mg + ritonavir (RTV) 100 mg + tenofovir (TDF) 300 mg + nucleoside of choice
  ATV , RTV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
- ATV 400 mg / SQV: ATV 400 mg + saquinavir (SQV) 1200 mg + TDF 300 mg + nucleoside of choice
  ATV, SQV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
- LPV / RTV: lopinavir (LPV)/RTV 400/100 mg + TDF 300 mg + nucleoside of choice
  LPV/RTV twice daily, TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
Period: Overall Study
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Started | 119 (120 randomized, 119 treated) | 110 (115 randomized, 110 treated) | 118 (123 randomized, 118 treated)
Discontinued Prior to Week 48 Visit | 26 | 29 | 13
Discontinued Between Weeks 48 and 96 | 26 | 27 | 30
Discontinued on or After Week 96 | 4 | 4 | 6
Completed | 63 (63 remained on treatment, 0 completed at Week 96) | 50 (50 remained on treatment, 0 completed at Week 96) | 69 (59 remained on treatment, 10 completed at Week 96)
Not Completed | 56 | 60 | 49
Not completed — Adverse Event | 10 | 9 | 9
Not completed — Death | 0 | 0 | 1
Not completed — Disease Progression / Relapse | 1 | 1 | 0
Not completed — Lost to Follow-up | 4 | 4 | 3
Not completed — Noncompliance | 6 | 7 | 6
Not completed — Protocol Violation While on Study | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 5 | 0
Not completed — Study Termination by Sponsor | 1 | 0 | 0
Not completed — Lack of Efficacy | 33 | 33 | 28

BASELINE CHARACTERISTICS:
Groups:
- ATV 300 mg / RTV: ATV 300 mg + RTV 100 mg + TDF 300 mg + nucleoside of choice
  ATV , RTV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
- ATV 400 mg / SQV: ATV 400 mg + SQV 1200 mg + TDF 300 mg + nucleoside of choice
  ATV, SQV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
- LPV / RTV: LPV/RTV 400/100 mg + TDF 300 mg + nucleoside of choice
  LPV/RTV twice daily, TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
- Total: Total of all reporting groups
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV | Total
Number analyzed (Participants) | 120 | 115 | 123 | 358
Age Continuous [Median (Full Range); unit: years] | 39 [24 to 71] | 41 [26 to 74] | 39 [25 to 72] | 40 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 27 | 77
  Male | 96 | 89 | 96 | 281
Race/Ethnicity, Customized [Number; unit: participants]
  White | 75 | 70 | 71 | 216
  Hispanic/Latino | 27 | 26 | 27 | 80
  Black | 18 | 16 | 21 | 55
  Other | 0 | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  South America | 56 | 55 | 54 | 165
  North America | 39 | 38 | 47 | 124
  Europe | 25 | 22 | 22 | 69
Acquired Immunodeficiency Virus (AIDS) [Number; unit: participants]
  Yes | 33 | 33 | 36 | 102
  No | 87 | 82 | 87 | 256
Intravenous (IV) Drug Use [Number; unit: participants]
  Yes | 8 | 7 | 8 | 23
  No | 112 | 108 | 115 | 335
Cluster of Differentiation 4 (CD4) cell count [Median (Full Range); unit: cells/mm^3] | 317 [40 to 1025] | 286 [42 to 1543] | 283 [14 to 1238] | 297 [14 to 1543]
Human Immunodeficiency Virus Ribonucleic Acid (HIV RNA) [Median (Full Range); unit: log10 c/mL] | 4.44 [2.60 to 5.88] | 4.42 [2.60 to 5.88] | 4.47 [2.60 to 5.88] | 4.45 [2.60 to 5.88]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in HIV Ribonucleic Acid (RNA) at Week 24
Time Frame: Baseline, Week 24
Population: Randomized participants; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
log10 c/mL | -1.86 (0.11) | -1.52 (0.13) | -1.89 (0.11)
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Non-Inferiority or Equivalence — The time-averaged difference (TAD) in the reduction of log10 HIV RNA levels from baseline through Week 24 was compared pairwise for each atazanavir regimen to the lopinavir/RTV regimen, and assessed using a two-sided 97.5% confidence interval. The primary efficacy analysis was to declare two treatment regimens similar if the upper limit of this 97.5% confidence interval for the difference (atazanavir-lopinavir/RTV) was less than 0.5 log10; Time-Averaged Difference = 0.14, 97.5% CI 2-sided [-0.09 to 0.37]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Time-Averaged Difference = 0.31, 97.5% CI 2-sided [0.07 to 0.55]

2. Secondary Outcome: Mean Change From Baseline in HIV RNA at Week 2
Time Frame: Baseline, Week 2
Population: Treated participants, as-randomized (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
log10 c/mL | -1.18 (0.06) | -1.14 (0.07) | -1.30 (0.06)
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Treatment Difference = 0.13, 95% CI 2-sided [-0.04 to 0.30]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Treatment Difference = 0.17, 95% CI 2-sided [-0.01 to 0.35]

3. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (Limit of Quantification [LOQ] = 400 c/mL) at Week 24 (Overall and by Protease Inhibitor [PI] Sensitivity)
Description: Number of participants with a >=0.5 log10 decrease in HIV RNA from baseline or HIV RNA < 400 c/mL at Week 24, by their baseline phenotypic sensitivity to their randomized PI.
Time Frame: Baseline, Week 24
Population: Number of Participants Analyzed=Randomized participants; as-randomized population (refers to the treatment regimen assigned at randomization); n=number of evaluable (overall, PI sensitive, PI resistant) participants.
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants
  Overall (n=120, 115, 123) | 95 | 74 | 93
  PI Sensitive (n=88, 83, 88) | 79 | 58 | 72
  PI Resistant (n=32, 30, 33) | 16 | 15 | 19

4. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (LOQ = 400 c/mL) at Week 48, (Overall and by PI Sensitivity)
Description: Number of participants with a >=0.5 log10 decrease in HIV RNA from baseline or HIV RNA < 400 c/mL at Week 48, by their baseline phenotypic sensitivity to their randomized PI.
Time Frame: Baseline, Week 48
Population: Number of Participants Analyzed=Randomized participants; as-randomized population (refers to the treatment regimen assigned at randomization).n=number of evaluable (overall, PI sensitive, PI resistant) participants.
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants
  Overall (n=120, 115, 123) | 77 | 60 | 84
  PI Sensitive (n=88, 84, 88) | 65 | 52 | 67
  PI Resistant (n=32, 30, 33) | 12 | 7 | 16

5. Primary Outcome: Mean Change From Baseline in HIV RNA at Week 48
Time Frame: Baseline, Week 48
Population: Randomized participants; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
log10 c/mL | -1.93 (0.12) | -1.55 (0.14) | -1.87 (0.13)
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Time-Averaged Difference = 0.13, 97.5% CI 2-sided [-0.12 to 0.39]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Time-Averaged Distance = 0.33, 97.5% CI 2-sided [0.07 to 0.60]

6. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (LOQ = 400 c/mL) at Week 96
Description: Number of participants with a >=0.5 log10 decrease in HIV RNA from baseline or HIV RNA < 400 c/mL at Week 96.
Time Frame: Baseline, Week 96
Population: Observed case analysis: Randomized participants (while on initial regimen--completers censored) with baseline and on-study measurement.
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | LPV / RTV
Number analyzed (Participants) | 120 | 113
participants | 61 | 58
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Randomized participants; Test type: Superiority or Other; Difference estimate = -0.5, 95% CI 2-sided [-13.3 to 12.3] — ATV 300/RTV - LPV/RTV

7. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (LOQ = 50 c/mL) at Week 24
Time Frame: Week 24
Population: Randomized participants; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants | 95 | 74 | 93
Statistical Analysis 1: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = 3.6, 95% CI 2-sided [-7.0 to 14.1]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -11.3, 95% CI 2-sided [-22.9 to 0.4]

8. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (LOQ = 50 c/mL) at Week 24, by PI Sensitivity
Description: Number of participants with a >=0.5 log10 decrease in HIV RNA from baseline or HIV RNA < 50 c/mL at Week 24, by their baseline phenotypic sensitivity to their randomized PI.
Time Frame: Baseline, Week 24
Population: As there were multiple efficacy algorithms run and multiple subsets analyzed, it was decided to only use LOQ < 50 on the primary endpoint, and to run LOQ<400 for subsets such as baseline PI sensitivity.
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (LOQ = 50 c/mL) at Week 48
Time Frame: Week 48
Population: Randomized participants; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
Participants | 76 | 60 | 84
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -5.0, 95% CI 2-sided [-16.9 to 7.0]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -16.1, 95% CI 2-sided [-28.5 to -3.7]

10. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (LOQ = 50 c/mL) at Week 48, by PI Sensitivity
Description: Number of participants with a >=0.5 log10 decrease in HIV RNA from baseline or HIV RNA < 50 c/mL at Week 48, by their baseline phenotypic sensitivity to their randomized PI.
Time Frame: Baseline, Week 48
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Participants Achieving Virologic Half Log Suppression (LOQ = 50 c/mL) at Week 96
Time Frame: Week 96
Population: Randomized participants while on initial regimen (completers censored).
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg / RTV | LPV / RTV
Number analyzed (Participants) | 120 | 113
Participants | 61 | 57
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = 0.4, 95% CI 2-sided [-12.5 to 13.2] — ATV 300/RTV - LPV/RTV

12. Secondary Outcome: Participants Achieving Treatment Response (LOQ = 400 c/mL) Without Prior Failure at Week 24
Description: Treatment Response = confirmed suppression to LOQ (400 c/mL). The Algorithm for Treatment Response Without Prior Failure (TRPWF) = participants staying in response at the analysis timepoint without having an intervening, confirmed rebound.
Time Frame: Week 24
Population: Randomized participants while on initial regimen Randomized participants, (completers censored).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants | 76 | 50 | 74
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = 3.2, 95% CI 2-sided [-9.1 to 15.4]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -16.7, 95% CI 2-sided [-29.4 to -4.0]

13. Secondary Outcome: Participants Achieving Treatment Response (LOQ = 400 c/mL) Without Prior Failure at Week 48
Description: as for outcome 12
Time Frame: Week 48
Population: Randomized participants, as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants | 64 | 42 | 67
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -1.1, 95% CI 2-sided [-13.7 to 11.4]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -17.9, 95% CI 2-sided [-30.6 to -5.3]

14. Secondary Outcome: Participants Achieving Treatment Response (LOQ = 400 c/mL) Without Prior Failure at Week 96
Description: as for outcome 12
Time Frame: Week 96
Population: Randomized participants while on initial regimen (completers censored).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | LPV / RTV
Number analyzed (Participants) | 120 | 116
participants | 52 | 53
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Chi-squared, Corrected; Difference Estimate = -2.4, 95% CI 2-sided [-15.0 to 10.3] — ATV 300/RTV - LPV/RTV

15. Secondary Outcome: Participants Achieving Treatment Response (LOQ = 50 c/mL) Without Prior Failure at Week 24
Description: Treatment Response = confirmed suppression to LOQ (50 c/mL). The Algorithm for Treatment Response Without Prior Failure (TRPWF) = participants staying in response at the analysis timepoint without having an intervening, confirmed rebound.
Time Frame: Week 24
Population: Randomized participants, as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants | 46 | 25 | 50
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -2.3, 95% CI 2-sided [-14.6 to 10.0]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -18.9, 95% CI 2-sided [-30.7 to -7.1]

16. Secondary Outcome: Participants Achieving Treatment Response (LOQ = 50 c/mL) Without Prior Failure at Week 48
Description: as for outcome 15
Time Frame: Week 48
Population: Randomized participantsRandomized participants while on initial regimen (completers censored).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants | 43 | 28 | 52
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -6.4, 95% CI 2-sided [-18.7 to 5.8]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Difference Estimate = -17.9, 95% CI 2-sided [-29.9 to -5.9]

17. Secondary Outcome: Participants Achieving Treatment Response (LOQ = 50 c/mL) Without Prior Failure at Week 96
Description: as for outcome 15
Time Frame: Week 96
Population: Randomized participants while on initial regimen (completers censored)
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | LPV / RTV
Number analyzed (Participants) | 120 | 118
participants | 38 | 41

18. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: Randomized participantsRandomized participants while on initial regimen (completers censored).
Measure: Mean (Standard Error); unit: cells/mm3
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
cells/mm3 | 83 (14.0) | 59 (11.8) | 90 (15.3)
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Time-Averaged Difference = -18.4, 97.5% CI 2-sided [-44.3 to 7.5]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Time-Averaged Difference = -44.9, 97.5% CI 2-sided [-74.5 to -15.3]

19. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Randomized participants while on initial regimen (completers censored).
Measure: Mean (Standard Error); unit: cells/mm3
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
cells/mm3 | 110 (22.9) | 72 (19.7) | 121 (20.1)
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Test type: Superiority or Other; Time-Averaged Difference = -17.5, 97.5% CI 2-sided [-45.6 to 10.6]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Test type: Superiority or Other; Time-Averaged Difference = -47.6, 97.5% CI 2-sided [-79.2 to -16.1]

20. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline, Week 96
Population: Randomized participants (while on initial regimen) with evaluation at time point
Measure: Mean (Standard Error); unit: cells/mm3
Arm/Group | ATV 300 mg / RTV | LPV / RTV
Number analyzed (Participants) | 60 | 60
cells/mm3 | 122 (26.3) | 154 (24.2)

21. Secondary Outcome: Correlation of ATV Minimum Plasma Concentration (Cmin), Inhibitory Quotient (IQ), and Number of Protease Inhibitor (PI) Mutations at Baseline With HIV RNA Change From Baseline at Week 24
Description: Pearson correlations of the Cmin (trough plasma concentration), IQ (the ratio of Cmin of ATV to HIV IC50), and Number of baseline PI Mutations with HIV RNA change from baseline at Week 24 were explored.
Time Frame: Baseline, Week 24
Population: Week 24: Participants with evaluable PK measurements
Measure: Number; unit: Pearson Correlation Coefficient
Groups:
- ATV 300 mg / RTV: ATV 300 mg + RTV 100 mg + TDF 300 mg + nucleoside of choice treated participants (HIV RNA change from baseline [log10 c/mL] Mean [SE] = -1.91 [0.19])
- ATV 400 mg / SQV: ATV 400 mg + SQV 1200 mg + TDF 300 mg + nucleoside of choice treated participants (HIV RNA change from baseline [log10 c/mL] Mean [SE] = -1.57 [0.3])
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 40 | 23
Pearson Correlation Coefficient
  ATV Cmin | -0.056 | 0.254
  IQ (<10; >=10) | -0.391 | -0.081
  # of PI Mutations at baseline (<4; >=4) | 0.306 | 0.437
Statistical Analysis 1: Comparison: ATV 300 mg / RTV; Correlation between IQ (<10; >=10) of ATV 300 mg / RTV and HIV RNA; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P-value was based on a t-distribution
Statistical Analysis 2: Comparison: ATV 400 mg / SQV; Correlation between number of PI Mutations at baseline (<4; >=4) of ATV 400 mg / SQV and HIV RNA; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P-value was based on a t-distribution

22. Secondary Outcome: Correlation of ATV Minimum Plasma Concentration (Cmin), Inhibitory Quotient (IQ), and Number of Protease Inhibitor (PI) Mutations at Baseline With HIV RNA Change From Baseline at Week 48
Description: Pearson correlations of the Cmin (trough plasma concentration), IQ (the ratio of Cmin of ATV to HIV IC50), and Number of baseline PI Mutations with HIV RNA change from baseline at Week 48 were explored.
Time Frame: Baseline, Week 48
Population: Formal population PK/PD analysis was not performed due to difficulties in correlating time of blood sample collection with drug administration, and inability to apply the PK model generated with data obtained from healthy subjects due to newly observed differences in exposure to atazanavir between HIV-infected participants and healthy participants.
Measure: Number; unit: Pearson Correlation Coefficient
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Correlation of ATV Minimum Plasma Concentration (Cmin) Inhibitory Quotient (IQ), and Number of PI Mutations at Baseline and CD4 Cell Count Change From Baseline at Week 24
Description: Pearson correlations of the Cmin (trough plasma concentration), IQ (the ratio of Cmin of ATV to HIV IC50), and Number of baseline PI Mutations with CD4 cell count change from baseline at Week 24 were explored.
Time Frame: Baseline, Week 24
Population: Participants with evaluable PK measurements, as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: Pearson Correlation Coefficient
Groups:
- ATV 300 mg / RTV: ATV 300 mg + RTV 100 mg + TDF 300 mg + nucleoside of choice treated participants (CD4 Cell Count Change from Baseline [cells/mm3] Mean [SE] = 80 [21])
- ATV 400 mg / SQV: ATV 400 mg + SQV 1200 mg + TDF 300 mg + nucleoside of choice treated participants (HIV RNA change from baseline [log10 c/mL] Mean [SE] = 56 [20])
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 40 | 23
Pearson Correlation Coefficient
  ATV Cmin | 0.37 | -0.21
  IQ (<10; >=10) | 0.376 | 0.105
  # of PI Mutations at baseline (<4; >=4) | -0.395 | -0.227
Statistical Analysis 1: Comparison: ATV 300 mg / RTV; Correlation between ATV Cmin of ATV 300 mg / RTV and CD4 Cell Count; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P-value was based on a t-distribution
Statistical Analysis 2: Comparison: ATV 300 mg / RTV; Correlation between IQ (<10; >=10) of ATV 300 mg / RTV and CD4 Cell Count; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P-value was based on a t-distribution
Statistical Analysis 3: Comparison: ATV 300 mg / RTV; Correlation between # of PI Mutations at baseline (<4; >=4) of ATV 300 mg / RTV and CD4 Cell Count; Test type: Superiority or Other; p < 0.05, t-test, 1 sided — P-value was based on a t-distribution

24. Secondary Outcome: Correlation of ATV Minimum Plasma Concentration (Cmin) Inhibitory Quotient (IQ), and Number of PI Mutations at Baseline and CD4 Cell Count Change From Baseline at Week 48
Description: Pearson correlations of the Cmin (trough plasma concentration), IQ (the ratio of Cmin of ATV to HIV IC50), and Number of baseline PI Mutations with CD4 cell count change from baseline at Week 48 were explored.
Time Frame: Baseline, Week 48
Population: as for outcome 22
Measure: Number; unit: Pearson Correlation Coefficient
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Lipid Mean Percent Change From Baseline at Week 24
Description: Mean percent change in total cholesterol, high density lipoprotein (HDL) cholesterol, fasting low density lipoprotein (LDL) cholesterol, and fasting triglycerides.
Time Frame: Baseline, Week 24
Population: Treated Participants, Last Observation Carried Forward (LOCF), as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: percent change
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
percent change
  Total Cholesterol | -8 | -9 | 3
  High Density Lipoprotein (HDL) Cholesterol | -7 | -1 | 0
  Fasting Low Density Lipoprotein (LDL) Cholesterol | -10 | -11 | -4
  Fasting Triglycerides | -2 | -14 | 31
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Total Cholesterol; Test type: Superiority or Other; Difference Estimate = -10.9, 95% CI 2-sided [-15.5 to -6.0]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Total Cholesterol; Test type: Superiority or Other; Difference Estimate = -12.4, 95% CI 2-sided [-16.9 to -7.6]
Statistical Analysis 3: Comparison: ATV 300 mg / RTV vs LPV / RTV; HDL cholesterol; Test type: Superiority or Other; Difference Estimate = -6.7, 95% CI 2-sided [-13.6 to 0.7]
Statistical Analysis 4: Comparison: ATV 400 mg / SQV vs LPV / RTV; HDL Cholesterol; Test type: Superiority or Other; Difference Estimate = -1.0, 95% CI 2-sided [-9.3 to 8.1]
Statistical Analysis 5: Comparison: ATV 300 mg / RTV vs LPV / RTV; Fasting LDL Cholesterol; Test type: Superiority or Other; Difference Estimate = -6.8, 95% CI 2-sided [-15.6 to 3.0]
Statistical Analysis 6: Comparison: ATV 400 mg / SQV vs LPV / RTV; Fasting LDL Cholesterol; Test type: Superiority or Other; Difference Estimate = -7.3, 95% CI 2-sided [-15.5 to 1.8]
Statistical Analysis 7: Comparison: ATV 300 mg / RTV vs LPV / RTV; Fasting Triglycerides; Test type: Superiority or Other; Difference Estimate = -24.9, 95% CI 2-sided [-35.0 to -13.2]
Statistical Analysis 8: Comparison: ATV 400 mg / SQV vs LPV / RTV; Fasting Triglycerides; Test type: Superiority or Other; Difference Estimate = -34.2, 95% CI 2-sided [-43.4 to -23.4]

26. Secondary Outcome: Lipid Mean Percent Change From Baseline at Week 48
Description: as for outcome 25
Time Frame: Week 48
Population: Treated Participants, Last Observation Carried Forward (LOCF); as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: percent change in lipid values
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
percent change in lipid values
  Total Cholesterol | -8 | -4 | 6
  HDL Cholesterol | -7 | 4 | 2
  Fasting LDL Cholesterol | -10 | -3 | 1
  Fasting Triglycerides | -4 | -14 | 30
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Total Cholesterol; Test type: Superiority or Other; Difference Estimate = -12.1, 95% CI 2-sided [-17.0 to -7.2]
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; Total Cholesterol; Test type: Superiority or Other; Difference Estimate = -12.0, 95% CI 2-sided [-17.4 to -6.5]
Statistical Analysis 3: Comparison: ATV 300 mg / RTV vs LPV / RTV; HDL Cholesterol; Test type: Superiority or Other; Difference Estimate = -4.4, 95% CI 2-sided [-12.4 to 3.5]
Statistical Analysis 4: Comparison: ATV 400 mg / SQV vs LPV / RTV; HDL Cholesterol; Test type: Superiority or Other; DIfference Estimate = -0.8, 95% CI 2-sided [-11.0 to 9.3]
Statistical Analysis 5: Comparison: ATV 300 mg / RTV vs LPV / RTV; Fasting LDL CHolesterol; Test type: Superiority or Other; Difference Estimate = -8.9, 95% CI 2-sided [-19.0 to 1.2]
Statistical Analysis 6: Comparison: ATV 400 mg / SQV vs LPV / RTV; Fasting LDL Cholesterol; Test type: Superiority or Other; Difference Estimate = -7.4, 95% CI 2-sided [-17.7 to 3.0]
Statistical Analysis 7: Comparison: ATV 300 mg / RTV vs LPV / RTV; Fasting Triglycerides; Test type: Superiority or Other; Difference Estimate = -29.6, 95% CI 2-sided [-41.6 to -17.7]
Statistical Analysis 8: Comparison: ATV 400 mg / SQV vs LPV / RTV; Fasting Triglycerides; Test type: Superiority or Other; Difference Estimate = -38.4, 95% CI 2-sided [-49.7 to -27.1]

27. Secondary Outcome: Lipid Mean Percent Change From Baseline at Week 96, Observed Values
Description: as for outcome 25
Time Frame: Week 96
Population: Treated Participants; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: percent change in lipid values
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
percent change in lipid values
  Total Cholesterol (n=60, 46, 54) | -7 | -1 | 9
  HDL Cholesterol (n=60, 46, 54) | -5 | 3 | 7
  Fasting LDL Cholesterol (n=52, 39, 43) | -11 | -7 | 1
  Fasting Triglycerides (n=52, 40, 43) | -2 | 4 | 30
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; Observed values, Total Cholesterol; Test type: Superiority or Other; Difference Estimate = -14.4, 95% CI 2-sided [-20.1 to -8.3] — ATV 300/RTV - LPV/RTV
Statistical Analysis 2: Comparison: ATV 400 mg / SQV vs LPV / RTV; observed values, total cholesterol; Test type: Superiority or Other; Difference Estimate = -9.0, 95% CI 2-sided [-16.1 to -1.3] — ATV 400/SQV - LPV/RTV
Statistical Analysis 3: Comparison: ATV 300 mg / RTV vs LPV / RTV; observed values, HDL cholesterol; Test type: Superiority or Other; Difference Estimate = -11.0, 95% CI 2-sided [-19.9 to -1.2] — ATV 300/RTV - LPV/RTV
Statistical Analysis 4: Comparison: ATV 400 mg / SQV vs LPV / RTV; Observed values, HDL cholesterol; Test type: Superiority or Other; Difference Estimate = -4.1, 95% CI 2-sided [-14.0 to 7.0] — ATV 400/SQV - LPV/RTV
Statistical Analysis 5: Comparison: ATV 300 mg / RTV vs LPV / RTV; observed cases, fasting LDL; Test type: Superiority or Other; Difference Estimate = -12.7, 95% CI 2-sided [-22.3 to -1.8] — ATV 300/RTV - LPV/RTV
Statistical Analysis 6: Comparison: ATV 400 mg / SQV vs LPV / RTV; Observed Cases, Fasting LDL cholesterol; Test type: Superiority or Other; Difference Estimate = -7.9, 95% CI 2-sided [-19.0 to 4.8] — ATV 400/SQV - LPV/RTV
Statistical Analysis 7: Comparison: ATV 300 mg / RTV vs LPV / RTV; observed cases, fasting triglycerides; Test type: Superiority or Other; Difference Estimate = -24.8, 95% CI 2-sided [-38.6 to -8.0] — ATV 300/RTV - LPV/RTV
Statistical Analysis 8: Comparison: ATV 400 mg / SQV vs LPV / RTV; observed cases, fasting triglycerides; Test type: Superiority or Other; Difference Estimate = -19.8, 95% CI 2-sided [-36.5 to 1.3] — ATV 400/SQV - LPV/RTV

28. Secondary Outcome: Deaths, Serious Adverse Events (SAEs), and Adverse Events (AEs) Through Week 48
Description: AE=any new untoward medical occurrence/worsening of a pre-existing medical condition regardless of causal relationship. SAE=any untoward medical occurrence at any dose that: results in death; is life-threatening; requires/prolongs inpatient hospitalization; results in persistent/significant disability; is cancer; is congenital anomaly/birth defect; results in drug dependency/abuse; is an important medical event.
Time Frame: From Enrollment through Week 48
Population: Randomized participants for Deaths and SAEs; treated participants for all others; as-randomized population (refers to the treatment regimen assigned at randomization). In addition, of the 213 screen failures (not randomized), there were 4 subjects who had an SAE; these are not included in the table below.
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 120 | 115 | 123
participants
  Deaths (n = 120, 115, 123) | 0 | 1 | 1
  AEs leading to discontinuation (n = 119, 110, 118) | 6 | 8 | 5
  SAEs (n = 120, 115, 123) | 12 | 14 | 11
  AEs, grades 1-4 (n = 119, 110, 118) | 97 | 93 | 103
  AEs, grades 3-4 (n = 119, 110, 118) | 11 | 18 | 12

29. Secondary Outcome: Most Common AEs and AEs of Interest Through Week 48
Description: Prespecified AEs of interest included jaundice, ocular icterus, and hyperbilirubinemia.
Time Frame: From Enrollment to Week 48
Population: Treated participants; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
participants
  Diarrhea (Most Common) | 25 | 29 | 54
  Headache (Most Common) | 21 | 24 | 18
  Nausea (Most Common) | 19 | 24 | 15
  Jaundice (AE of Interest) | 19 | 6 | 0
  Ocular Icterus (AE of Interest) | 13 | 3 | 0
  Hyperbilirubinemia (AE of Interest) | 24 | 8 | 1

30. Secondary Outcome: Fasting Glucose Mean Change From Baseline at Week 24
Time Frame: Baseline, Week 24
Population: Treated Participants with evaluation at time point; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 104 | 87 | 99
mg/dL | 0 (1.6) | -3 (1.8) | 0 (1.4)

31. Secondary Outcome: Fasting Glucose Mean Change From Baseline at Week 48
Time Frame: Week 48
Population: as for outcome 30
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 115 | 108 | 112
mg/dL | 4 (3.6) | -1 (1.6) | 1 (1.5)

32. Secondary Outcome: Grade 3/4 Laboratory Abnormalities Through Week 48
Description: Common Terminology Criteria for Adverse Events v3.0 (CTCAE) Grades:1=Mild, 2=Moderate, 3=Severe, 4=Life-threatening/disabling, 5=Death. Abnormal values: absolute neutrophil count: ≥500 to <750/mm3 (grade 3), <500/mm3 (grade 4); platelets: 20,000-49,999/mm3 (grade 3), <20,000/mm3 or diffuse petechiae (grade 4); alanine transaminase (ALT): 5.1-10 x upper limit of normal (ULN; grade 3), >10 x ULN (grade 4); aspartate transaminase (AST): 5.1-10 x ULN (grade 3), >10 x ULN (grade 4); bilirubin: 2.6-5 x ULN (grade 3), >5 x ULN (grade 4).
Time Frame: From Enrollment to Week 48
Population: Evaluable treated participants; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 108 | 118
participants
  Neutrophil Reduction | 8 | 8 | 10
  Platelet Reduction | 2 | 4 | 3
  ALT Elevation | 5 | 4 | 4
  AST Elevation | 4 | 2 | 4
  Total Bilirubin Elevation | 58 | 22 | 1

33. Secondary Outcome: Fridericia-corrected QT (QTcF) Interval and Change From Baseline by Analysis Time Point
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. The QT interval was corrected for heart rate using Fridericia's (QTcF) formula.
Time Frame: Baseline, Week 4 predose, 2-3 hours postdose, 6-12 hours postdose, Week 12, Week 24, Week 48
Population: Treated participants; as-randomized population (refers to the treatment regimen assigned at randomization). n=number of participants evaluated at timepoint
Measure: Mean (Standard Error); unit: msec
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
msec
  Baseline Mean (n=119, 110, 118) | 390 (1.9) | 387 (2.2) | 390 (1.9)
  Mean Change at Week 4 predose (n=117, 104, 110) | -3 (1.6) | 1 (1.9) | -2 (1.7)
  Mean Change Wk 4 2-3 hrs postdose (n=113,102,106) | -2 (1.6) | -3 (2.0) | -7 (1.9)
  Mean Change Wk 4 6-12 hrs postdose (n=112,101,105) | -4 (1.7) | -1 (1.9) | -8 (1.8)
  Mean Change at Week 12 (n=110, 97, 107) | 2 (1.6) | 3 (2.0) | 2 (1.6)
  Mean Change at Week 24 (n=108, 92, 109) | 1 (1.8) | 3 (2.2) | 2 (1.8)
  Mean Change at Week 48 (n=89, 75, 97) | -1 (1.8) | -1 (2.1) | 0 (2.0)

34. Secondary Outcome: PR Interval and Change From Baseline by Analysis Time Point
Description: The PR interval is measured from the beginning of the P wave to the beginning of the QRS complex, and reflects the time the electrical impulse takes to travel from the sinus node through the atrioventricular (AV) node and entering the ventricles. The PR interval is therefore a good estimate of AV node function.
Time Frame: Baseline, Week 4 predose, 2-3 hours postdose, 6-12 hours postdose, Week 12, Week 24, Week 48
Population: as for outcome 33
Measure: Mean (Standard Error); unit: msec
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
msec
  Baseline Mean (n=119, 110, 118) | 153 (1.7) | 155 (1.9) | 154 (1.7)
  Mean Change at Week 4 predose (n=117, 104, 110) | 4 (1.2) | 9 (1.6) | 3 (1.4)
  Mean Change Wk 4 2-3 hrs postdose (n=113,102,106) | 1 (1.3) | 6 (1.6) | 1 (1.7)
  Mean Change Wk 4 6-12 hrs postdose (n=112,101,105) | 2 (1.4) | 6 (1.7) | 2 (1.5)
  Mean Change at Week 12 (n=110, 97, 107) | 5 (1.6) | 7 (1.7) | 8 (1.4)
  Mean Change at Week 24 (n=108, 92, 109) | 2 (1.3) | 7 (1.7) | 5 (1.6)
  Mean Change at Week 48 (n=89, 75, 97) | 0 (1.5) | 2 (1.9) | 4 (1.7)

35. Secondary Outcome: Adherence to Regimen Though Week 48 Based on MACS the Multicenter AIDS Cohort Study (MACS) Adherence Questionnaire
Description: The MACS adherence questionnaire asks patients how many medication doses they missed during the previous day, 2 days, 3 days and 4 days. Drug-specific questions included adherence with dose and frequency. Adherence was defined as taking all doses and numbers of pills as prescribed for each medication. This strict adherence cut-off was based on the guidelines stating that anything less than excellent adherence may result in a virus breakthrough and development of resistance.
Time Frame: Baseline, Week 24, Week 48
Population: Number of Participants Analyzed=treated participants; as-randomized population (refers to the treatment regimen assigned at randomization); n=subset of treated participants (Given the language limitation, a subset of the AI424045 population was included in the MACS adherence analysis.)
Measure: Number; unit: participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 40 | 33 | 48
participants
  Adherent at Baseline (n=27, 25, 33) | 12 | 10 | 18
  Adherent at Week 24 (n=18, 11, 25) | 10 | 5 | 23
  Adherent at Week 48 (n=11, 4, 20) | 8 | 2 | 13

36. Secondary Outcome: Mean Score of European Quality of Life-5 Dimensions (EQ-5D) Health Index Score at Baseline, Mid-Study (Week 24), and Final (Week 48)
Description: The EQ-5D is a 5-item questionnaire to assess health-related quality of life in 5 health dimensions (mobility, self-care, usual activity, pain/discomfort, anxiety/depression) are scored on a 3-level scale: no problems (1), some problems (2), extreme problems (3). Using a standard algorithm, responses are summarized into a single score, the EQ-5D Health Index Score (HIS), which ranges between 1 (representing perfect health) and 0 (representing the worst imaginable health state or death). The smallest coefficient of change is 0.03.
Time Frame: Baseline, Week 24, Week 48
Population: Treated participants; as-randomized population (refers to the treatment regimen assigned at randomization). n=number of participants evaluated with EQ-5D at given time point.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
units on a scale
  Baseline (n=99, 86, 100) | 0.83 (0.02) | 0.85 (0.02) | 0.86 (0.02)
  Mid-Study (n=103, 83, 95) | 0.87 (0.02) | 0.86 (0.02) | 0.89 (0.01)
  Final (n=93, 84, 96) | 0.84 (0.02) | 0.85 (0.03) | 0.88 (0.02)

37. Secondary Outcome: Mean Score of European Quality of Life-5 Dimensions (EQ-5D) Visual Analog Scale (VAS) at Baseline, Mid-Study (Week 24), and Final (Week 48)
Description: The EQ-5D has a Visual Analog Scale (VAS), which is a feeling thermometer-like scale with a range between 0 and 100. Patients are required to draw a line from a box on the VAS scale to an actual mark on the thermometer-like scale that corresponds with a number that reflects their self-assessed health status at the time they are completing the questionnaire. Higher VAS scores indicate better overall health. There is no minimum clinically important difference reported in the literature for VAS.
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 36
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 119 | 110 | 118
units on a scale
  Baseline (n=98, 85, 101) | 81.33 (1.63) | 81.72 (1.77) | 81.52 (1.53)
  Mid-Study (n=102, 83, 97) | 84.89 (1.65) | 83.34 (1.89) | 85.09 (1.55)
  Final (n=95, 81, 96) | 82.77 (1.72) | 85.80 (1.64) | 86.16 (1.36)

38. Primary Outcome: Mean Change From Baseline in HIV RNA at Week 96
Time Frame: Baseline, Week 96
Population: Randomized participants while on initial regimen
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | ATV 300 mg / RTV | LPV / RTV
Number analyzed (Participants) | 64 | 65
log10 c/mL | -2.29 (0.121) | -2.08 (0.151)
Statistical Analysis 1: Comparison: ATV 300 mg / RTV vs LPV / RTV; overall; Test type: Superiority or Other; time-averaged difference = 0.14, 97.5% CI 2-sided [-0.13 to 0.41] — ATV 300/RTV - LPV/RTV
Statistical Analysis 2: Comparison: ATV 300 mg / RTV vs LPV / RTV; last observation carried forward; Test type: Superiority or Other; time-averaged difference = 0.11, 97.5% CI 2-sided [-0.16 to 0.38] — ATV 300/RTV - LPV/RTV

39. Secondary Outcome: Number of Participants Utilizing Resources for Managing Lipid Elevation
Description: Participants' overall resource utilization for managing lipid elevation that includes the management of side effects of lipid lowering medications, such as those due to drug interactions.
Time Frame: Baseline, Week 24, Week 48
Population: Although the intent of this planned analysis was to provide a model of economic value for Lipid Management, a different approach was taken to create this model which did not require data from this trial, and thus this analysis was not done.
Measure: Number; unit: Participants
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV | LPV / RTV
Number analyzed (Participants) | 0 | 0 | 0

40. Secondary Outcome: Mean ATV, RTV and SQV Minimum Concentration (Cmin) Values
Description: The minimum or "trough" concentration (Cmin) of a drug observed after its administration and just prior to the administration of a subsequent dose.
Time Frame: collected at the pre-dose time point after receiving atazanavir for at least four weeks
Population: Participants with evaluable Cmins; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 40 | 23
ng/mL
  ATV (n=40,23) | 719.53 (82.81) | 312.01 (145.31)
  RTV (n=40,0) | 154.83 (39.31) | NA (NA) — No participants were analyzed in this cohort for RTV because they did not take this drug.
  SQV (n=0,19) | NA (NA) — No participants were analyzed in this cohort for SQV because they did not take this drug. | 52.15 (16.89)

41. Secondary Outcome: HIV IC50 at Week 24
Description: IC50: inhibitory concentration of drug required to reduce viral replication by 50%.
Time Frame: Week 24
Population: Participants with evaluable IC50 measurements; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 40 | 21
ng/mL | 17.83 (4.04) | 22.84 (11.65)

42. Secondary Outcome: Inhibitory Quotient at Week 24
Description: Inhibitory quotient is a measure of drug exposure and susceptibility in an individual. The IQ is typically calculated as the ratio of Cmin to HIV IC50.
Time Frame: Baseline, Week 24
Population: Participants with evaluable IQ measurements (ie, must have both Cmin and IC50 measurements); as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: ratio
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 40 | 21
ratio | 136.94 (24.33) | 25.04 (13.33)

43. Secondary Outcome: Inhibitory Quotient at Week 48
Description: as for outcome 42
Time Frame: Baseline, Week 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: ratio
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: HIV RNA Level - Treated Subjects With Evaluable Cmins at Week 24
Description: Week 24 HIV RNA level and change from baseline were summarized for treated subjects with evaluable Cmins.
Time Frame: Baseline, Week 24
Population: Participants with evaluable Cmins; as-randomized population (refers to the treatment regimen assigned at randomization).
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 40 | 23
log10 c/mL
  Baseline Values | 4.53 (0.13) | 4.41 (0.13)
  Week 24 Values | 2.62 (0.19) | 2.83 (0.25)
  Change from Baseline at Week 24 | -1.91 (0.19) | -1.57 (0.29)

45. Secondary Outcome: HIV RNA Level - Treated Subjects With Evaluable Cmins at Week 48
Description: Week 24 HIV RNA level and change from baseline were summarized for treated subjects with evaluable Cmins.
Time Frame: Baseline, Week 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: log10 c/mL
Arm/Group | ATV 300 mg / RTV | ATV 400 mg / SQV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The AE data below represents data from start of study in November 2001 through the last locked database of the study, 18 November 2009.
Groups:
- ATV300/RTV: atazanavir (ATV) 300 mg + ritonavir (RTV) 100 mg + tenofovir (TDF) 300 mg + nucleoside of choice ATV , RTV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
- ATV400/SQV: ATV 400 mg + saquinavir (SQV) 1200 mg + TDF 300 mg + nucleoside of choice ATV, SQV, and TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
- LPV/RTV: lopinavir (LPV)/RTV 400/100 mg + TDF 300 mg + nucleoside of choice LPV/RTV twice daily, TDF once daily, nucleoside per label 48 Weeks and then for as long as subject is in need of therapy through study
Arm/Group | ATV300/RTV | ATV400/SQV | LPV/RTV
Serious Adverse Events (participants affected / at risk) | 22/119 | 22/110 | 19/118
Other Adverse Events (participants affected / at risk) | 101/119 | 95/110 | 104/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATV300/RTV (N=119) | ATV400/SQV (N=110) | LPV/RTV (N=118)
GLAUCOMA (Eye disorders) | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 0 | 1 | 1
PERICARDITIS (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 0 | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0
ANEURYSM (Vascular disorders) | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 0 | 0 | 1
DRUG ABUSE (Psychiatric disorders) | 0 | 1 | 1
ALCOHOL ABUSE (Psychiatric disorders) | 0 | 1 | 0
DRUG DEPENDENCE (Psychiatric disorders) | 1 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 1 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 | 0 | 2
HYPERSENSITIVITY (Immune system disorders) | 1 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 1 | 0
TENSION HEADACHE (Nervous system disorders) | 0 | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 2
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 1
PANCREATITIS (Gastrointestinal disorders) | 1 | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 2 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0
UROSEPSIS (Infections and infestations) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
ABSCESS LIMB (Infections and infestations) | 0 | 1 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 2
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0
NEUROSYPHILIS (Infections and infestations) | 0 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 0
CRYPTOCOCCOSIS (Infections and infestations) | 1 | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 2 | 0 | 0
MENINGITIS TUBERCULOUS (Infections and infestations) | 0 | 0 | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 1
RENAL TUBULAR ACIDOSIS (Renal and urinary disorders) | 0 | 0 | 1
HOSPITALISATION (Surgical and medical procedures) | 0 | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERLACTACIDAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 1
PROSTATITIS (Reproductive system and breast disorders) | 0 | 1 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 2 | 0
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 | 0 | 1
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 0 | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 2 | 0 | 2
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
CYST (General disorders) | 0 | 1 | 0
CHILLS (General disorders) | 0 | 1 | 0
MALAISE (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 1 | 1 | 2
CHEST PAIN (General disorders) | 0 | 1 | 1
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
CARCINOID TUMOUR OF THE GASTROINTESTINAL TRACT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATV300/RTV (N=119) | ATV400/SQV (N=110) | LPV/RTV (N=118)
OCULAR ICTERUS (Eye disorders) | 13 | 4 | 0
LIPASE INCREASED (Investigations) | 8 | 2 | 8
WEIGHT DECREASED (Investigations) | 10 | 9 | 13
BLOOD BILIRUBIN INCREASED (Investigations) | 11 | 4 | 1
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 7 | 2 | 9
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 2 | 6
ANXIETY (Psychiatric disorders) | 8 | 9 | 4
INSOMNIA (Psychiatric disorders) | 12 | 6 | 10
DEPRESSION (Psychiatric disorders) | 12 | 11 | 14
JAUNDICE (Hepatobiliary disorders) | 19 | 7 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 23 | 8 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 6 | 2
HEADACHE (Nervous system disorders) | 23 | 28 | 22
DIZZINESS (Nervous system disorders) | 7 | 9 | 7
PARAESTHESIA (Nervous system disorders) | 5 | 5 | 10
HYPOAESTHESIA (Nervous system disorders) | 2 | 2 | 8
NEUROPATHY PERIPHERAL (Nervous system disorders) | 5 | 4 | 7
NAUSEA (Gastrointestinal disorders) | 23 | 30 | 18
VOMITING (Gastrointestinal disorders) | 16 | 17 | 12
DIARRHOEA (Gastrointestinal disorders) | 30 | 34 | 63
DYSPEPSIA (Gastrointestinal disorders) | 7 | 10 | 6
GASTRITIS (Gastrointestinal disorders) | 1 | 6 | 1
FLATULENCE (Gastrointestinal disorders) | 6 | 8 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 12 | 10
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 6 | 8 | 8
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 16 | 7
INFLUENZA (Infections and infestations) | 20 | 17 | 14
PNEUMONIA (Infections and infestations) | 6 | 5 | 3
SINUSITIS (Infections and infestations) | 15 | 14 | 19
BRONCHITIS (Infections and infestations) | 13 | 12 | 17
PHARYNGITIS (Infections and infestations) | 8 | 7 | 7
GASTROENTERITIS (Infections and infestations) | 2 | 4 | 7
NASOPHARYNGITIS (Infections and infestations) | 17 | 13 | 19
URINARY TRACT INFECTION (Infections and infestations) | 10 | 9 | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 5 | 14
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 | 12 | 12
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 8 | 6 | 8
RASH (Skin and subcutaneous tissue disorders) | 7 | 10 | 12
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 7 | 6
LIPOATROPHY (Skin and subcutaneous tissue disorders) | 2 | 6 | 5
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 9 | 10 | 11
MYALGIA (Musculoskeletal and connective tissue disorders) | 12 | 6 | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 15 | 13 | 13
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 | 10 | 7
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 7 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 17
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 11
FATIGUE (General disorders) | 9 | 10 | 10
PYREXIA (General disorders) | 19 | 9 | 10
ASTHENIA (General disorders) | 7 | 7 | 9
OEDEMA PERIPHERAL (General disorders) | 2 | 2 | 6
INFLUENZA LIKE ILLNESS (General disorders) | 8 | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.